CLINICAL TRIAL: NCT04216511
Title: Clinic Validation of Autoantibody Panel for Lung Cancer Diagnosis in Chinese Population
Brief Title: Early Cancer Detection Test - Lung Cancer China
Acronym: ECLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bai Chunxue (Other)
Collaborators: Gene Tech (Shanghai) Company Limited (Unknown)
Responsible Party: Sponsor-Investigator, Bai Chunxue, Chairman, Chinese Alliance Against Lung Cancer
Organization: Chinese Alliance Against Lung Cancer (Other)
Other Study IDs: CAALC-007-EarlyCDT Lung China
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Tumor Autoantibody; Early Detection; Indeterminate Pulmonary Nodule
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum or plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-Lung Cancer: Patients with definite lung cancer diagnosis
  Interventions: Diagnostic Test: Tumor autoantibody detection
- Control: Either patients with benign pulmonary nodule, or healthy individuals without pulmonary nodule but with risk factors to develop lung cancer matched to lung cancer group
  Interventions: Diagnostic Test: Tumor autoantibody detection

INTERVENTIONS:
Diagnostic Test: Tumor autoantibody detection — Level of a set of autoantibodies potentially relative with lung cancer will be tested for each of the participants.

SUMMARY:
Lung cancer is the most common cancer in China from both incidence and mortality rate point of view, with significantly lower 5-year survival rate than average. Early detection is the recognized solution. LDCT is more and more popular accepted as an effective screening methodology but leads to numerous indeterminate pulmonary nodules for physicians to distinguish too. The value of autoantibody test in risk assessing of IPNs as well as early detection of lung cancer in high risk population has been demonstrated in clinical practice and trial but mainly in Caucasian. Purpose of this study is to understand the sensitivity, specificity and accuracy of candidate autoantibodies, and consequently explore the autoantibody combination with best clinical performance in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or above.
* Individuals complying with either of the following

  1. diagnosed as lung cancer (histopathologically confirmed);
  2. diagnosed as benign pulmonary nodule (confirmed by pathology or by follow-up based on 2018 Chinese Consensus on Pulmonary Nodule Diagnosis and Treatment);
  3. without pulmonary nodule but with lung cancer risk factor, age & gender matched recruited lung cancer patients.
* Participant is willing and able to provide necessary information required in CRF.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* History of any cancer;
* Lung cancer patient who received or is receiving any treatment, including but not limited to surgery, radiotherapy, chemotherapy, targeted therapy and immunotherapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with lung cancer, benign pulmonary nodule or identified as at-risk healthy volunteer in participating hospitals of this study, from the recruitment starting date, till the end of the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Autoantibody panel with best clinical performance in Chinese population | Oct.30, 2020
  The combination which can achieve best sensitivity at 90% specificity, and its sensitivity, accuracy and PPV.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxue Bai, MD, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai
  - Henan Province People's Hospital, Zhengzhou